CLINICAL TRIAL: NCT06405009
Title: A Nomogram for Predicting Occult Omental Metastasis in Patients With Gastric Cancer
Brief Title: Prediction Model of Occult Omental Metastasis in Patients With Gastric Cancer
Status: Recruiting | Type: Observational
Sponsor: Northern Jiangsu People's Hospital (Other)
Responsible Party: Principal Investigator, Daorong Wang, Clinical Professor, Northern Jiangsu People's Hospital
Other Study IDs: NorthernJiangsu003
Record Dates: First submitted 2024-04-22; First posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Gastric Cancer; Omental Metastasis
MeSH Terms: conditions — Stomach Neoplasms | interventions — Risk Factors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with omental metastases
  Interventions: Other: Without any intervention, we only divided gastric cancer patients into two groups based on postoperative pathology, and analyzed their basic characteristics and risk factors
- patients without omental metastases
  Interventions: Other: Without any intervention, we only divided gastric cancer patients into two groups based on postoperative pathology, and analyzed their basic characteristics and risk factors

INTERVENTIONS:
Other: Without any intervention, we only divided gastric cancer patients into two groups based on postoperative pathology, and analyzed their basic characteristics and risk factors — Without any intervention, we only divided gastric cancer patients into two groups based on postoperative pathology, and analyzed their basic characteristics and risk factors

SUMMARY:
A complete omentectomy is typically recommended during radical total gastrectomy for gastric cancer, though its impact on survival remains unclear. This study aimed to assess the frequency and risk factors of metastases in the greater omentum in gastric cancer patients undergoing gastrectomy. It will involve a single prospective cohort of consecutive patients who underwent total gastrectomy with complete en bloc omentectomy and modified D2 lymphadenectomy. Post-surgery, the omentum will dissect from the gastrectomy specimen beyond the gastroepiploic vessels and examine separately for pathological assessment. The primary outcome will focus on the detection of omental metastases.

ELIGIBILITY:
Inclusion Criteria:

1. pathological confirmation of gastric cancer
2. eligibility for surgical intervention
3. undergoing first rectal cancer surgery
4. acquisition of written informed consent from patients and their families
5. no history of hypertrophic scar or allergic predispositions

Exclusion Criteria:

1. absence of postoperative pathology of the omentum
2. diagnosis of multiple primary malignancies
3. intraoperative discovery of widespread implant metastases within the abdominal cavity
4. severe comorbidities

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: It included consecutive patients with a primary gastric adenocarcinoma (cT1-4N0-3M0) in whom a potentially curative total gastrectomy could be performed.
Sampling Method: Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2024-04-22 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
patients with omental metastases | up to 2 weeks after gastric cancer surgery
  After the operation, the postoperative pathological examination of the patient indicated the presence of omental metastases
patients without omental metastases | up to 2 weeks after gastric cancer surgery
  After surgery, pathological examination confirmed no omental metastases

CONTACTS AND LOCATIONS:
Locations (1):
- Yifan Cheng, Yangzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No